CLINICAL TRIAL: NCT04711083
Title: Correlation Between Nocturnal Oxygen Desaturation and Glycemic Control in Diabetic Patients With Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr Shoukri, Assistant Professor of pulmonary medicine, Ain Shams University
Other Study IDs: OPO10-18
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Obstructive Sleep Apnea; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus, Type 2 | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: overnight pulse oximetry — Wrist worn Overnight oximetry was performed using portable Nonin 2500 (Nonin Medical Inc., USA) pulse oximeters. The test was explained to the subjects and their caregiver by experienced health-care staff from the sleep unit. The recording was done at home and started just before going to bed and ended on awakening; the recommended duration was a minimum of 5 h and a maximum of 7 h. The awake SpO2, mean SpO2. The data were analysed to calculate the overnight minimum SpO2, mean SpO2, dip frequency (defined as a fall in SpO2 of > 4%), the percentage of oximetry sleep time spent with a SpO2 of < 90%, and the total oximetry time. Recordings were classified as "normal" (< 4.9 desaturation events an hour), "equivocal" (5 to 14.9 desaturation events an hour), or "abnormal" (> 15 desaturation events an hour) according to the severity and pattern of nocturnal desaturation observed .
  Other Names: polysomnography

SUMMARY:
Nocturnal reduction in blood oxygen is expected independently associated with the development of worsened glycemic control in individuals with type 2 diabetes mellitus.

The aim of the present study is to assess the correlation between nocturnal oxygen desaturation assessed by overnight pulse oximetry and glycemic control in diabetic patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
Introduction:

Obstructive sleep apnea syndrome (OSAS) is a prevalent illness showing a heterogeneous symptom presentation, which ranges from low clinical suspicion to evident limitations in the quality of life. The main reasons for this variability relate to its potential association with major concomitant diseases, which include diabetes and a variety of cardiovascular pathologies. (1).

Also, OSA is a known risk factor for many comorbid disorders, causing resistance to conventional treatments and increasing the risk of mortality, which multiplies health care expenditures and even though the distribution of comorbidities differs between men and women, their effect progressively increases with OSA severity (2,3) Occurrence of apneic events and Reduction in blood oxygen and elevations in blood carbon dioxide are sensed by chemoreceptors in the brain and carotid bodies, which trigger brief microarousals and result in sleep fragmentation (4).

Nocturnal reduction in blood oxygen has also been independently associated with the development of worsened glycemic control in individuals with type 2 diabetes (4).

Aim of the work:

to assess the correlation between nocturnal oxygen desaturation assessed by overnight pulse oximetry and glycemic control in diabetic patients with obstructive sleep apnea.

Material and Methods:

This study will be conducted on all patients referred for evaluation of sleep related breathing disorders. All Medical files were reviewed. Data collected included .full medical history, demographics, measurements of weight and height, body mass index in kg/m2, neck circumference (NC), Epworth Sleepiness Scale (ESS) scores, measurements of overnight pulse oximetryglyceminc control (measurement of glycated HB, fasting and 2h postprandial blood sugar)The diagnosis that was concluded after a polysomnography study.

ELIGIBILITY:
Inclusion Criteria:

* All patient swith type 2 diabetes, referred for evaluation of sleep related breathing disorder

Exclusion Criteria:

* Patients less than 18 years old and Patients receiving treatment for sleep related breathing disorders were excluded

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients 18 years old or above, with type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
correlation between nocturnal oxygen desaturation and glycemic control | 1 year
  measurements of blood glucose control and nocturnal oxygen level.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
results of noxturnal oximetry, patients demographics.